CLINICAL TRIAL: NCT07089992
Title: URSa-1: A Minibasket Study of Pembrolizumab in Ultra-Rare Sarcomas
Brief Title: A Study of Pembrolizumab in People With Ultra-Rare Sarcomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-165
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma
Keywords: Pleomorphic liposarcoma; PEComa (perivascular epithelial cell tumor); Epithelioid sarcoma; CIC-rearranged sarcoma; SEF/LGFMS: Sclerosing epithelioid fibrosarcoma - low grade fibromyxoid sarcoma; Ultra-Rare Sarcomas; Pembrolizumab; 25-165
MeSH Terms: conditions — Sarcoma; Liposarcoma; Perivascular Epithelioid Cell Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pleomorphic liposarcoma (Experimental): Pembrolizumab Q 6 weeks IV infusion
  Interventions: Drug: Pembrolizumab
- PEComa (perivascular epithelial cell tumor) (Experimental): Pembrolizumab Q 6 weeks IV infusion
  Interventions: Drug: Pembrolizumab
- Epithelioid sarcoma (Experimental): Pembrolizumab Q 6 weeks IV infusion
  Interventions: Drug: Pembrolizumab
- CIC-rearranged sarcoma (Experimental): Pembrolizumab Q 6 weeks IV infusion
  Interventions: Drug: Pembrolizumab
- Sclerosing epithelioid fibrosarcoma - low grade fibromyxoid sarcoma (Experimental): Pembrolizumab Q 6 weeks IV infusion
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Q 6 weeks IV infusion Day 1 of each 6-week cycle, up to 8 doses

SUMMARY:
The purpose of the study is to find out if pembrolizumab is a useful treatment that causes few or mild side effects in people with ultra-rare sarcoma. The researchers will also study how the immune system responds to the study treatment.

Pembrolizumab is a type of drug called a PD-1 inhibitor. It is designed to block a protein called programmed cell death protein 1 (PD-1) that usually acts as a "brake" on the immune system. Blocking this protein is like releasing the brakes, so that the immune system can target cancer cells and destroy them.

ELIGIBILITY:
Inclusion:

* Patients must have pathologically confirmed diagnosis of one of the following:

  1. Pleomorphic liposarcoma
  2. PEComa (perivascular epithelial cell tumor)
  3. Epithelioid sarcoma
  4. CIC-rearranged sarcoma
  5. SEF/LGFMS: Sclerosing epithelioid fibrosarcoma - low grade fibromyxoid sarcoma
* Molecular characterization of the tumor, if available, will be recorded. If no such molecular data are available, note as such.
* Patient should have recurrent or metastatic disease not judged to be curable with other means
* Patients must have progressed (in the opinion of the treating investigator) following the most recent line of therapy. The reason for this progression must be documented, employing tumor measurements when available.
* Definition of Measurable Disease

  * Measurable disease as per RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions for a minimum of 3 months after completion of such therapy
  * Patients with treated brain metastases are eligible if follow up brain imaging after CNS-directed therapy shows no evidence of progression at least 4 weeks after the completion of therapy as shown by follow up imaging before study screening
  * One to 3 prior lines of therapy are permitted (including neoadjuvant/adjuvant or metastatic/recurrent disease)
  * Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible. Patients with alopecia and other toxicities considered clinically nonsignificant and/or stable on supportive therapy, as determined by the investigator, are also permitted on study.
  * Administration of killed vaccines is allowed
* Age ≥ 18 years of age.
* ECOG Performance Status 0-1 (Karnofsky 70-100)
* Required organ function (specimens to be collected within 14 days of the start of the study intervention)

  * Adequate hematologic function, defined as:

    * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm^3
    * Platelets ≥ 100,000 cells/mm^3
    * Hemoglobin ≥ 9 g/dl
  * Adequate renal function defined, as:

    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert disease who have bilirubin level ≤ 3 x ULN may be enrolled)
    * AST and ALT ≤3 x institutional ULN
  * Adequate cardiac function, defined as: class II or better New York Heart Association (NYHA) Functional Classification.
  * For patients with known HIV, HBV, and/or HCV infection [HIV, HBV, and HCV testing do not need to be performed as part of the study; the below language provides guidelines for inclusivity of patients with known HIV, HBV, and/or HCV infection]:

    * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months and CD4+ T cell count of at least 350 cell/mm3 are eligible for this trial.
    * HIV-infected patients with a history of either Kaposi sarcoma or Castleman disease are excluded from this study
    * HIV-infected patients must not have had an AIDS defining opportunistic infection within the past 12 months
  * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

Exclusion:

* No prior diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drug.
* No other active malignancy, other than breast or prostate cancer stable for at least 6 months on hormonal therapy, or CLL Rai stage 0. Cancer in situ will not be considered an active malignancy.
* No active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid)
* No prior (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Must have adequately recovered from major surgery (at least 4 weeks), without ongoing surgical complications. Patients should have had any minor procedures (e.g. port placement, percutaneous nephrostomy) at least 2 weeks prior to the first day of treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's ability to cooperate with the requirements of the study participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* No known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Not pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* No prior allogenic tissue/solid organ transplant.
* Patients with documented leptomeningeal disease are excluded from study, even if treated.
* No prior systemic anti-cancer therapy including investigational agents within 4 weeks, 2 weeks for kinase inhibitors or intravenous chemotherapy, prior to starting therapy on study
* No investigational agent(s) administration or use of investigational device within 4 weeks prior to study intervention administration.
* No prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
* No prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* No live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention.
* No known bleeding diathesis (e.g. hemophilia, DIC)
* No active infection requiring systemic therapy
* No history of allergic reaction to the study agent(s), compounds of similar chemical or biologic composition to the study agent (s) (or any of its excipients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 12 weeks
  iRECIST, which is based on RECIST 1.1

SECONDARY OUTCOMES:
Toxicity assessment | 2 years
  NCI CTCAE Version 5, Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org